CLINICAL TRIAL: NCT04419441
Title: Retrospective, Multicentric, Observational Study to Evaluate the Efficacy and Safety of the Combination of an Immune Checkpoint Inhibitor (ICI) and Radiotherapy (RT) in Patients With Relapsed/Refractory (R/R) Classical Hodgkin Lymphoma (cHL)
Brief Title: Immune Checkpoint Inhibitors and Radiotherapy in Relapsed/Refractory Hodgkin Lymphoma
Acronym: ICI-RT-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Maggiore Di Trieste (Other)
Responsible Party: Principal Investigator, Francesco Zaja, Professor, Ospedale Maggiore Di Trieste
Other Study IDs: ICI-RT-01
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Hodgkin Lymphoma; Immune Checkpoint Inhibitor; Radiotherapy
MeSH Terms: conditions — Hodgkin Disease | interventions — Immune Checkpoint Inhibitors; Radiotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- treated patients: patients with relapsed/refractory Hodgkin lymphoma who received a treatment with the combination of radiotherapy and an immune checkpoint inhibitor
  Interventions: Drug: Immune checkpoint inhibitor

INTERVENTIONS:
Drug: Immune checkpoint inhibitor — concomitant administration of radiotherapy and immune checkpoint inhibitor
  Other Names: radiotherapy

SUMMARY:
This is an observational retrospective study to investigate the efficacy and safety of the treatment with an immune checkpoint inhibitor (nivolumab or pembrolizumab) in combination with radiotherapy in patients with relapsed/refractory classical Hodgkin lymphoma.

DETAILED DESCRIPTION:
In patients with relapsed/refractory Hodgkin lymphoma, treatment with immune checkpoint inhibitors (ICIs), nivolumab and pembrolizumab, leads to 20-30% of complete remission (CR) rate. This means that for the majority of patients a consolidation strategy is usually offered, in order to reduce relapse rate.

Strategies to improve CR rates should therefore be implemented, including combination treatments. In solid tumors, the combination of ICIs and radiotherapy led to higher response rates without mjor toxicity concerns. Radiotherapy is an effective therapeutic option already used in Hodgkin lymphoma patients, also in the setting of relapsed/refractory disease. In his observational study we aim to evaluate the efficacy and safety of ICIs and radiotherapy administered in combination in patients with relapsed/refractory Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* diagnosis of classical Hodgkin lymphoma, treated with one immune checkpoint inhibitor (ICI) (nivolumab or pembrolizumab), as per label indication
* having received a concomitant radiotherapy, as per clinical need (persistence of localized disease, bulky disease, other reasons). "Concomitant" radiotherapy means a treatment received during the administration of ICI, or during the 8 weeks that precede or follow the start or the end of the treatment with ICI

Exclusion Criteria:

* Having received a treatment with an ICI and radiotherapy not "concomitant", according to the abovementioned definition
* Having received any other anti-lymphoma treatments during the same period of time
* Patients who have not been evaluated by CT-PET or CT at the end of the combination therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients with relapsed/refractory Hodgkin lymphoma treated in referral centers for haematology
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) rate measured according to Lugano and Lyric criteria by CT-PET (positron emission tomography / computer tomography) or CT (computer tomography) scan | up to 2 months after the end of ICI or 3 months after the end of RT

SECONDARY OUTCOMES:
overall response rate (ORR) measured according to Lugano and Lyric criteria by CT-PET or CT scan | up to 2 months after the end of ICI or 3 months after the end of RT
progression-free survival (PFS) measured according to Cheson 2007 response criteria | from the start of the treatment until the date of documented progression or date of death from any cause, assessed up to 5 years
safety profile assessed by monitoring adverse events (AEs) and serious adverse events (SAEs) according to CTCAE v. 4.0 | through study completion, for an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zaja, Professor, Principal Investigator — SC Ematologia Ospedale Maggiore Trieste
Locations (1):
- SC Ematologia Ospedale Maggiore, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided
it is not yet known if there will be a plan to make IPD available

REFERENCES:
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Cheson BD, Ansell S, Schwartz L, Gordon LI, Advani R, Jacene HA, Hoos A, Barrington SF, Armand P. Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy. Blood. 2016 Nov 24;128(21):2489-2496. doi: 10.1182/blood-2016-05-718528. Epub 2016 Aug 29. PMID 27574190
- [Background] Armand P, Engert A, Younes A, Fanale M, Santoro A, Zinzani PL, Timmerman JM, Collins GP, Ramchandren R, Cohen JB, De Boer JP, Kuruvilla J, Savage KJ, Trneny M, Shipp MA, Kato K, Sumbul A, Farsaci B, Ansell SM. Nivolumab for Relapsed/Refractory Classic Hodgkin Lymphoma After Failure of Autologous Hematopoietic Cell Transplantation: Extended Follow-Up of the Multicohort Single-Arm Phase II CheckMate 205 Trial. J Clin Oncol. 2018 May 10;36(14):1428-1439. doi: 10.1200/JCO.2017.76.0793. Epub 2018 Mar 27. PMID 29584546
- [Background] Chen R, Zinzani PL, Lee HJ, Armand P, Johnson NA, Brice P, Radford J, Ribrag V, Molin D, Vassilakopoulos TP, Tomita A, von Tresckow B, Shipp MA, Lin J, Kim E, Nahar A, Balakumaran A, Moskowitz CH. Pembrolizumab in relapsed or refractory Hodgkin lymphoma: 2-year follow-up of KEYNOTE-087. Blood. 2019 Oct 3;134(14):1144-1153. doi: 10.1182/blood.2019000324. Epub 2019 Aug 13. PMID 31409671
- [Background] Constine LS, Yahalom J, Ng AK, Hodgson DC, Wirth A, Milgrom SA, Mikhaeel NG, Eich HT, Illidge T, Ricardi U, Dieckmann K, Moskowitz CH, Advani R, Mauch PM, Specht L, Hoppe RT. The Role of Radiation Therapy in Patients With Relapsed or Refractory Hodgkin Lymphoma: Guidelines From the International Lymphoma Radiation Oncology Group. Int J Radiat Oncol Biol Phys. 2018 Apr 1;100(5):1100-1118. doi: 10.1016/j.ijrobp.2018.01.011. Epub 2018 Jan 9. PMID 29722655
- [Background] Chen L, Douglass J, Kleinberg L, Ye X, Marciscano AE, Forde PM, Brahmer J, Lipson E, Sharfman W, Hammers H, Naidoo J, Bettegowda C, Lim M, Redmond KJ. Concurrent Immune Checkpoint Inhibitors and Stereotactic Radiosurgery for Brain Metastases in Non-Small Cell Lung Cancer, Melanoma, and Renal Cell Carcinoma. Int J Radiat Oncol Biol Phys. 2018 Mar 15;100(4):916-925. doi: 10.1016/j.ijrobp.2017.11.041. Epub 2017 Dec 5. PMID 29485071